CLINICAL TRIAL: NCT00853476
Title: The Standard Concentration of Morphine as a Positive Control for Intradermal Skin Test
Status: Completed | Type: Observational
Sponsor: Chulalongkorn University (Other)
Responsible Party: Jettanong Klaewsongkram, MD, Chulalongkorn University
Other Study IDs: Chula-ARC 001/09
Record Dates: First submitted 2009-02-27; First posted 2009-03-02 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2011-02

CONDITIONS: Intradermal Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to compare skin reactivity results between morphine and histamine as a positive control agents in intradermal skin test.

DETAILED DESCRIPTION:
Histamine hydrochloride and different concentrations of morphine sulfate will be intradermally injected and wheal diameter size will be comparatively measured between 15-30 minutes' time points after the test.

ELIGIBILITY:
Inclusion Criteria:

* age 18-60 years old

Exclusion Criteria:

* immunodeficiency state
* cancer
* severe skin diseases
* severe medical illnesses
* malnutrition
* uncontrolled asthma
* pregnancy
* received oral or systemic corticosteroid within 1 month before this study
* receiving immunosuppressive agents
* taken antihistamine within 3 days before this study
* taking beta-blocker
* previous history of immunotherapy
* have hypersensitivity reaction to morphine/opiates

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adult Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2009-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Wheal diameter from morphine skin test at different concentrations compared to standard histamine between 15-30 minutes after skin test | 30 minutes

SECONDARY OUTCOMES:
Side effects | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jettanong Klaewsongkram, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand